CLINICAL TRIAL: NCT04101695
Title: Hemodynamic Response of Anodal Transcranial Direct Current Stimulation (tDCS) Over the Cerebellar Hemisphere in Healthy Subjects: A Pilot Trial
Brief Title: Hemodynamic Response of Anodal Transcranial Direct Current Stimulation Over the Cerebellar Hemisphere in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won-Seok Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1908-558-004
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Transcranial Direct Current Stimulation; Functional Near Infrared Spectroscopy
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS- washout period- anodal tDCS (Active Comparator): Ybrain tDCS System (Ybrain, Korea) is used. Anode of tDCS is placed over right cerebellar hemisphere (3cm lateral from the occipital protuberance) and cathode over the on ipsilateral buccinator muscle.
  For Sham tDCS, total stimulation lasts 90 seconds: ramp up period of 30 seconds, stimultation for intensity of 2mA for 30 seconds, and ramp down period of 30 seconds. At least 7 days of washout period is in between two tDCS. For Anodal tDCS, 20 minutes of stimulation for intensity of 2mA.
  Interventions: Device: tDCS
- anodal tDCS- washout period- sham tDCS (Active Comparator): Ybrain tDCS System (Ybrain, Korea) is used. Anode of tDCS is placed over right cerebellar hemisphere (3cm lateral from the occipital protuberance) and cathode over the on ipsilateral buccinator muscle.
  For Anodal tDCS, 20 minutes of stimulation for intensity of 2mA. At least 7 days of washout period is in between two tDCS. For Sham tDCS, total stimulation lasts 90 seconds: ramp up period of 30 seconds, stimultation for intensity of 2mA for 30 seconds, and ramp down period of 30 seconds.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Ybrain tDCS System (Ybrain, Korea) is used for anodal stimulation of cerebellar hemisphere. Anode of tDCS is placed over right cerebellar hemisphere (3cm lateral from the occipital protuberance) and cathode over the on right buccinator muscle.

SUMMARY:
Upper extremity motor impairment is one of the major sequelae of stroke, resulting in limitation of activities of daily livings. Noninvasive neuromodulation is one of the therapies for motor recovery, which includes transcranial magnetic stimulation and transcranial direct current stimulation(tDCS). Anodal tDCS increases excitability and cathodal tDCS decreases excitability of neurons.

In systematic reviews, tDCS applied over primary motor cortex showed positive results on motor learning and improvements of hand fine motors. Recently, there has been trials of tDCS over cerebellum, considering the connectivity of primary motor cortex and cerebellum in motor controls. However, the results of these trials are yet contradictory, and the study using the functional near infrared spectroscopy to prove the effects of tDCS over distant area is lacking.

Therefore, in this study, we used functional near infrared spectroscopy (fNIRS) to observe the hemodynamic change of primary motor cortex when applying tDCS over cerebellum ascertain their connectivity.

In this crossover design, participants are randomly allocated to "sham tDCS-washout period-anodal tDCS group" or "anodal tDCS- washout period- sham tDCS group". The recording of fNIRS starts 3 minutes before the tDCS stimulation and continues throughout 20 minutes of stimulation, until 30 minutes after the stimulation cessation. After 7 days of washout period, second recording is done as the same protocol. Outcome measures are the changes of concentration of deoxyhemoglobin [deoxy-Hb] and oxyhemoglobin [oxy-Hb].

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 years or older
* No known brain disorders

Exclusion Criteria:

* Uncontrolled or unstalbe medical condition
* Pregnant
* Scalp problem which interferese with tDCS
* metals in the head (example: clip, coil), cochlear implants

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Changes of concentration of deoxyhemoglobin | comparison between sham and anodal tDCS (at least 7 days apart)
  detected by fNIRS and implies cortical metabolic changes
Changes of concentration of oxyhemoglobin | comparison between sham and anodal tDCS (at least 7 days apart)
  detected by fNIRS and implies cortical metabolic changes

CONTACTS AND LOCATIONS:
Overall Officials: Won-Seok Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Please Select, South Korea

IPD SHARING:
Plan to Share IPD: No
We are not planning to share the individual data publicly.